CLINICAL TRIAL: NCT01552200
Title: Performance Evaluation of the NaviAid™ G-Eye System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smart Medical Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: G-Eye 15501
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Colorectal Cancer; Polyp; Adenoma
Keywords: Colorectal Cancer; Polyp; Adenoma; Detection Rate; Colonoscopy; NaviAid™ G-Eye procedure; NaviAid™ G-Eye system; G-Eye procedure; G-Eye system
MeSH Terms: conditions — Colorectal Neoplasms; Polyps; Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A-Standard Colonoscopy, G-Eye procedure (Experimental): Standard Colonoscopy,G-Eye procedure
  Interventions: Procedure: Group A-Standard Colonoscopy, then NaviAid™ G-Eye procedure
- B- G-Eye procedure, Standard Colonoscopy (Active Comparator): G-Eye procedure,Standard Colonoscopy
  Interventions: Procedure: Group B-NaviAid™ G-Eye procedure, then Standard Colonoscopy

INTERVENTIONS:
Procedure: Group A-Standard Colonoscopy, then NaviAid™ G-Eye procedure — Standard Colonoscopy,NaviAid™ G-Eye procedure
  Arms: A-Standard Colonoscopy, G-Eye procedure
Procedure: Group B-NaviAid™ G-Eye procedure, then Standard Colonoscopy — G-Eye procedure, Standard Colonoscopy
  Arms: B- G-Eye procedure, Standard Colonoscopy

SUMMARY:
The purpose of this study is to compare the additional diagnostic yield obtained by performing NaviAid™ G-Eye procedure vs. the diagnostic yield obtained by performing standard colonoscopy procedure.

DETAILED DESCRIPTION:
Colonoscopy is the gold-standard method for CRC screening, as it enables detection and real-time removal of pre-cancerous polyps during the examination. It is well known that lesions are missed during routine colonoscopy.5 major reasons can be detailed for missing polyps during colonoscopy: polyps that are hidden behind folds, polyps that are masked by the colon's topography and natural folds, shallow polyps, unscreened portions of the colon (due to incomplete colonoscopy) and endoscope slippage. The NaviAid™ G-Eye system presents a unique concept that overcomes all 5 items listed above, providing an overall solution to the two endoscopy key challenges of limited detection/treatment yield and limited operation range.

The G-Eye endoscope comprises a standard endoscope onto which a unique balloon is permanently integrated, at its bending section. The NaviAid™ G-Eye may be used for performing controlled withdrawal and endoscope stabilization.

A major attribute of the NaviAid™ G-Eye system controlled withdrawal technique of the endoscope, with the balloon moderately inflated is to expand and stretch the intestinal lumen during endoscope withdrawal.

This is a multicenter, two-arm, randomized, open-label study intended to compare the additional diagnostic yield obtained by performing NaviAid™ G-Eye procedure vs. the diagnostic yield obtained by performing standard colonoscopy procedure.

Subjects will be randomized to one of two groups: Group A, the "Study Group," and Group B, the "Control Group."

Group A: Subjects will undergo a complete standard colonoscopy as the first procedure. Immediately after the standard colonoscopy procedure, a complete NaviAid™ G-Eye procedure will be performed by the same endoscopist.

Group B: Subjects will undergo a complete NaviAid™ G-Eye procedure as the first procedure. Immediately after the NaviAid™ G-Eye procedure, a complete standard colonoscopy will be performed by the same endoscopist.

ELIGIBILITY:
Inclusion Criteria:

* The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic workup;
* The patient is over 40 years old;
* The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

* Subjects with inflammatory bowel disease;
* Subjects with a personal history of polyposis syndrome;
* Subjects with suspected chronic stricture potentially precluding complete colonoscopy;
* Subjects with diverticulitis or toxic megacolon;
* Subjects with a history of radiation therapy to abdomen or pelvis;
* Pregnant or lactating female subjects;
* Subjects who are currently enrolled in another clinical investigation.
* Subjects with routine oral or parenteral use of anticoagulants
* Subjects with recent (within the last 3 mounts) coronary ischemia or CVA (stroke)
* Any patient condition deemed too risky for the study by the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
NaviAid™ G-Eye procedure adenoma detection rate compared to the standard colonoscopy procedure adenoma detection rate | Subjects will be followed during the study period (approximatly 3 hours) and follow up will be done within 48-72 hours following the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Erwin Santo, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center; Beny Shpak, MD, Principal Investigator — Laniado Hospital; Yael Kopelman, MD, Principal Investigator — Hadassah Medical Organization
Locations (4):
- St. Marienkrankenhaus Frankfurt, Frankfurt, Germany
- Israel (3):
  - Hadassah Medical Organization, Jerusalem
  - Laniado Hospital, Netanya
  - Tel Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Derived] Halpern Z, Gross SA, Gralnek IM, Shpak B, Pochapin M, Hoffman A, Mizrahi M, Rochberger YS, Moshkowitz M, Santo E, Melhem A, Grinshpon R, Pfefer J, Kiesslich R. Comparison of adenoma detection and miss rates between a novel balloon colonoscope and standard colonoscopy: a randomized tandem study. Endoscopy. 2015 Mar;47(3):238-44. doi: 10.1055/s-0034-1391437. Epub 2015 Feb 17. PMID 25704662